CLINICAL TRIAL: NCT05840211
Title: A Randomized, Open-label, Phase 3 Study of Sacituzumab Govitecan Versus Treatment of Physician's Choice in Patients With Hormone Receptor-Positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2-) (HER2 IHC0 or HER2-low [IHC 1+, IHC 2+/ISH-]) Inoperable, Locally Advanced, or Metastatic Breast Cancer and Have Received Endocrine Therapy
Brief Title: Study of Sacituzumab Govitecan Versus Treatment of Physician's Choice in Patients With Hormone Receptor-positive/Human Epidermal Growth Factor Receptor 2 Negative (HR+/HER2-) Metastatic Breast Cancer Who Have Received Endocrine Therapy
Acronym: ASCENT-07
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-598-6168; 2022-502593-17-00 (Other: European Medicines Agency); jRCT2061230032 (Other: Japan Registry of Clinical Trials); DOH-27-082023-6901 (Other: South African National Clinical Trials Registry); MOH_2023-07-17_012821 (Other: Israel Clinical Research Site); CTR20233370 (Registry Identifier: China: Drug Clinical Trial Registration and Information Disclosure Platform)
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Unresectable Metastatic Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan-hziy (SG) (Experimental): Participants will receive SG at a dose of 10 mg/kg infusion on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Treatment of Physician's Choice (TPC) (Active Comparator): Participants will receive TPC determined prior to randomization to 1 of the 3 allowed regimens:
  * paclitaxel 80 mg/m^2 over 1 hour (± 10 minutes) on Days 1, 8, and 15 of a 28-day cycle.
  * nab-Paclitaxel 100 mg/m^2 over 30 minutes (± 10 minutes) on Days 1, 8, and 15 of a 28-day cycle.
  * capecitabine at 1000-1250 mg/m^2 twice daily for 2 weeks followed by a 1-week rest period of a 21-day cycle.
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: Trodelvy™; GS-0132; IMMU-132
  Arms: Sacituzumab Govitecan-hziy (SG)
Drug: Paclitaxel — Administered intravenously
  Other Names: Taxol®
  Arms: Treatment of Physician's Choice (TPC)
Drug: Nab-paclitaxel — Administered intravenously
  Other Names: Abraxane®
  Arms: Treatment of Physician's Choice (TPC)
Drug: Capecitabine — Administered orally
  Other Names: Xeloda®
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
The goal of this clinical study is to see if sacituzumab govitecan-hziy (SG) can improve life spans of people with HR+/HER2- metastatic breast cancer and their tumor does not grow or spread when compared to currently available standard treatments, such as paclitaxel, nab-paclitaxel or capecitabine. The primary objective is to compare the effect of SG relative to the treatment of physician's choice (TPC) on progression-free survival (PFS).

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and give written informed consent.
* Must have adequate tumor tissue sample preferably from locally recurrent or metastatic site.
* Documented evidence of HR+ metastatic breast cancer (mBC) confirmed with the most recently available tumor biopsy preferably from a locally recurrent or metastatic site.
* Documented evidence of HER2- status.
* Documented PD by computed tomography (CT) or magnetic resonance imaging during or after the most recent therapy per RECIST v1.1 criteria.
* Candidate for the first chemotherapy in the locally advanced or metastatic setting.
* Eligible for capecitabine, nab-paclitaxel, or paclitaxel.
* Individuals must have at least one of the following:

  * Disease progression on at least 2 or more previous lines of endocrine therapy (ET) with or without a targeted therapy in the metastatic setting.

    * Disease recurrence while on the first 24 months of starting adjuvant ET will be considered a line of therapy; these individuals will only require 1 line of ET in the metastatic setting.
  * Disease progression within 6 months of starting first-line ET with or without a cyclin-dependent kinase (CDK) 4/6 inhibitor (if ineligible or if unable to access a CDK 4/6 inhibitor) in the metastatic setting.
  * Disease recurrence while on the first 24 months of starting adjuvant ET with CDK 4/6 inhibitor and if the individual is no longer a candidate for additional ET in the metastatic setting.
* Individuals may have received prior targeted therapies, including but not limited to PARP inhibitors (for those with germline BRCA1 or BRCA2 mutations), phosphatidylinositol 3-kinase (PI3K) inhibitors (for those with PIK3CA mutations), or mammalian target of rapamycin (mTOR) inhibitors. However, individuals can no longer be candidates for additional endocrine treatment with or without targeted therapies.
* Individuals with HIV must be on antiretroviral therapy (ART) and have a well-controlled HIV infection/disease.
* Demonstrates adequate organ function.
* Male individuals and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Key Exclusion Criteria:

* Progressive disease within 6 months of completing (neo)adjuvant chemotherapy.
* Locally advanced metastatic breast cancer (mBC) (Stage IIIc) in individuals who are candidates for curative intent therapy at the time of study enrollment.
* Current enrollment in another clinical study and use of any investigational device or drug (drugs not marketed for any indication) either within 5 half-lives or 28 days prior to randomization, whichever is longer.

  * Use of investigational drugs in the category of Selective Estrogen Receptor Degraders are acceptable if last dose was longer than 14 days prior to randomization.
* Received any prior treatment (including antibody-drug conjugate (ADC)) containing a chemotherapeutic agent targeting topoisomerase I.
* Received any prior treatment with a trophoblast cell-surface antigen 2 (Trop-2)-directed ADC.
* Have an active second malignancy.
* Have an active serious infection requiring antibiotics.
* Have active hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Individuals positive for human immunodeficiency virus type 1/2 (HIV-1 or -2) with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
* Have a positive serum pregnancy test or are breastfeeding for individuals who are assigned female at birth.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Up to approximately 29 months
  PFS is defined as time from date of randomization until the date of first objective progressive disease (PD) or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Until death, up to approximately 60 months
  OS is defined as the time from randomization until the date of death from any cause.
Objective Response Rate (ORR) as Assessed by BICR per RECIST Version 1.1 | Until progression, up to approximately 60 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.
Change from Baseline in the Physical Functioning Domain Using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Version 3.0 (EORTC QLQ-C30) at Week 16 | Baseline, Week 16
  The EORTC QLQ-C30 is composed of global health status/QoL scale; five functional domains (physical, role, emotional, cognitive, and social); three symptom domains (fatigue, nausea and vomiting, and pain); and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
  The Physical Functioning domain includes 5 questions in which participants will be asked to rate their overall health and overall quality of life as it relates to physical functioning during the past week on a scale from 1 (very poor) to 4 (excellent), with a higher score representing a high QoL.
Time to Deterioration in Version 3.0 EORTC-QLQ-C30 Scores | Up to approximately 60 months
  Time to deterioration from baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores. Scale scores range from 0-100. For functioning and global health status/QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden.
Progression Free Survival (PFS) as Assessed by Investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Until progression or death, up to approximately 60 months
  PFS is defined as time from date of randomization until the date of first objective progressive disease (PD) by investigator assessment according to RECIST v1.1 or death from any cause, whichever comes first.
Objective Response Rate (ORR) as Assessed by Investigator per RECIST Version 1.1 | Up to approximately 60 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.
Duration of Response (DOR) as Assessed by BICR and Investigator per RECIST Version 1.1 | Until progression or death, up to approximately 60 months
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of objective PD or death from any cause (whichever comes first).
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | First dose date up to 30 days post last dose, up to approximately 60 months
Percentage of Participants Experiencing Clinically Significant Laboratory and/or Vital Sign Abnormalities | First dose date up to 30 days post last dose, up to approximately 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (288):
- United States (30):
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Chandler, Arizona
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of California, San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Rocky Mountain Cancer Centers, LLP, Littleton, Colorado
  - Yale-New Haven Hospital-Yale Cancer Center, New Haven, Connecticut
  - Investigational Drug Services, AdventHealth Orlando, Altamonte Springs, Florida
  - Florida Cancer Specialists, Brooksville, Florida
  - Florida Cancer Specialist, Leesburg, Florida
  - Florida Cancer Specialist, St. Petersburg, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Georgia Cancer Specialist - Annex, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - The University of Kansas Hospital, Kansas City, Kansas
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - David C. Pratt Cancer Center, St Louis, Missouri
  - Astera Cancer Care, East Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - Magee-Womens of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - US Oncology Investigational Products Center (IPC), Fairfax, Virginia
  - US Oncology Investigational Products Center (IPC), Norfolk, Virginia
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
- Argentina (7):
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas de Mar del Plata, Buenos Aires
  - Instituto Alexander Fleming, C.a.b.a.
  - Hospital Alemán, CABA
  - Centro Privado de RMI Rio Cuarto S.A., Córdoba
  - Instituto de Oncología de Rosario, Rosario
  - CER San Juan Centro Polivalente de Asistencia e Investigación Clínica, San Juan
- Australia (10):
  - Royal Brisbane and Women's Hospital, Queensland, ME
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - GenesisCare North Shore (Oncology), St Leonards, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Austin Health, Melbourne, Victoria
  - Sunshine Hospital (Western Health), St Albans, Victoria
  - Breast Cancer Research Centre - WA, Nedlands, Western Australia
- Austria (4):
  - University Hospital Innsbruck, Innsbruck
  - Universitätsklinik für Innere Medizin 3 der PMU, Salzburg
  - Medizinische Universitat Wien, Univ. Klinik fur Innere Medizin I Klinische Abteilung fur Onkologie, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (5):
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Antwerp
  - AZ Klina, Brasschaat
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitaire Ziekenhuis Leuven, Leuven
  - CHU UCL Namur-Site STE. Elisabeth, Namur
- Brazil (20):
  - Hospital Haroldo Juaçaba - Instituto do Câncer do Ceará, Fortaleza
  - Hospital Araujo Jorge - Associacao de Combate ao Cancer em Goias, Goiânia
  - Oncosite - Centro de Pesquisa Clinica e Oncologia, Ijuí
  - Catarina Pesquisa Clinica, Itajaí
  - Oncoclinicas do Brasil Servicos Medicos AS, Minas Gerais
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal
  - CIONC-Centro Integrado de Oncologia de Curitiba, Paraana
  - Hospital Erasto Gaertner, Paraná
  - IMIP - Instituto de Medicina Integral Professor Fernando Figueira, Pernambuco
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Porto Alegre - HCPA, Porto Alegre
  - HGB - Hospital Giovanni Battista/Mãe de Deus Center, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Instituto Americas, Rio de Janeiro
  - Clínica de Oncologia de Porto Alegre Ltda - CLINIONCO, Rio Grande
  - Unidade de PesquisasClinicas em Oncologia - UPCO, Rio Grande
  - Instituto do Câncer - Hospital São Vicente de Paulo, Rio Grande
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Instituto Hemomed Oncologia e Hematologia, São Paulo
  - Clinica de pesquisa e centro de estudos em oncologia ginecológica e mamaria, São Paulo
- Canada (5):
  - BC Cancer - Kelowna, Kelowna
  - The Ottawa Hospital Cancer Centre, Ottawa
  - CHU de Québec-Université Laval, Hôpital du Saint-Sacrement, Québec
  - Humber River Hospital, Toronto
  - BC Cancer-Victoria, Victoria
- Chile (5):
  - Centro de Investigacion Clinica Bradford Hill, Recoleta
  - Centro del Cancer UC, Region Metropolitana
  - Centro de Oncología de Precisión (COP), Santiago Region
  - James Lind Centro de Investigacion del Cancer, Temuco
  - Oncocentro APYS, Viña del Mar
- China (29):
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Anhui
  - Peking University People's Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Cancer Hospital, Fujian
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - Sir Run Run Shaw Hospital,Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Heilongjiang
  - Jiangsu Province Hospital, Jiangsu
  - The First Affiliated Hospital of Soochow University, Jiangsu
  - The Nanchang Third Hospital, Jiangxi
  - The Second Hospital of Jilin University, Jilin Sheng
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - General Hospital of Ningxia Medical University, Ningxia Hui
  - The Affiliated Hospital Of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (7):
  - Fakultni Nemocnice Brno, Brno
  - Masaryk Memorial Cancer Institute, Brno
  - University Hospital Olomouc, Olomouc
  - Multiscan s.r.o, Pardubice
  - Charles General University Hospital, Prague, Prague
  - Fakultni nemocnice v Motole, Prague
  - Krajska nemocnice Tomase Bati Zlin, Zlín
- France (16):
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Clinique Francois Chenieux, Limoges
  - Ico René Gauducheau, Loire Atlantique
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Regional du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Hopital Privé des Cotes d'Armor, Plérin
  - Centre Jean Bernard Service d'Oncologie Médicale, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (14):
  - Universitaetsklinikum Freiburg, Klinik fuer Frauenheilkunde, Baden-Württemberg
  - University Hospital rechts der Isar Technical University of Munich, Bayern
  - Vivantes Klinikum am Urban, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Marienhospital Bottrop, Bottrop
  - Universitätsklinik Erlangen, Erlangen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Nationales Centrum für Tumorerkrankungen Heidelberg, Heidelberg
  - Universitätsklinikum Mannheim, Mannheim
  - LMU Klinikum der Universitat München, München
  - Universitatsklinikum Munster, Münster
  - Universitäts - Frauenklinik, Tübingen
- Greece (7):
  - Alexandra General Hospital, Athens
  - Attikon Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - Bioclinic of Thessaloniki, Thessaloniki
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
- Hong Kong (3):
  - Hong Kong Integrated Oncology Centre, Hong Kong
  - Prince of Wales Hospital, New Territories
  - Queen Mary Hospital, Pok Fu Lam
- Hungary (5):
  - Semmelweis Egyetem, Belgyogyaszati es Onkologiai Klinika, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Bács-Kiskun Varmegyei Oktatokorhaz, Onkaradiologiai Kozpont, Kecskemét
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz, Onkoradiologia, Nyíregyháza
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Israel (6):
  - Oncology Institute Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (17):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona AN
  - Centro di Riferimento Oncologico - IRCCS, Aviano
  - Humanitas Gavazzeni, Bergamo
  - ASST Papa Giovanni XXIII, Bergamo
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola, Bologna
  - Humanitas Istituto Clinico Catanese, Catania
  - Azienda Ospedaliera Mater Domini, Catanzaro
  - IRCCS Ospedale Policlinico San Martino, Genova GE
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS San Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Istituto Oncologico Veneto IOV, Padua
  - Irccs Crob, Rionero in Vulture
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (25):
  - Aichi Cancer Center Hospital, Aichi
  - Tohoku University Hospital, Aoba-ku
  - Juntendo University Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital, Chūōku
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Chūōku
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - Fukushima Medical University Hospital, Fukushima
  - Social Medical Corporation Hakuaikai Sagara Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - National Cancer Center Hospital East, Kashiwa
  - Saitama Cancer Center, Kitaadachi-gun
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Kyushu Cancer Center, Minamiku
  - Nagoya University Hospital, Nagoya
  - Hiroshima City Hiroshima Citizens Hospital, Nakaku
  - Hyogo Medical University Hospital, Nishinomiya-shi
  - Okayama University Hospital, Okayama
  - Gunma Prefectural Cancer Center, Ōta-ku
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku
  - Showa University Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Malaysia (4):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Institut Kanser Negara, Putrajaya
- Mexico (7):
  - Centro de Investigacion y Avances Medicos Especializados, Cancún
  - COI Centro Oncologico Internacional S.A.P.I. de C.V., Mexico City
  - FUCAM, México
  - Hospital Universitario Dr. José Eleuterio González, Monterrey
  - Clinica Integral Internacional de Oncologia S de RL de CV, Puebla City
  - Centro Medico Zambrano Hellion, San Pedro Garza García
  - Centro de Atención e Investigación Clínica en Oncología, Yucatán
- Poland (6):
  - Copemicus Podmiot Leczniczy Wojewodzkie Centrum Okologii w Gdansku, Gdansk
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie Sp. z.o.o, Krakow
  - Instytut MSF Sp. z o.o., Lodz
  - Wojewodzki Szpital Specjalistyczny lm. Stefana Kardynala Wyszynsklego SPZOZ w Lublinie, Lublin
  - LUX MED Onkologia Sp. Zo.o., Warsaw
  - Maria Sklodowska - Curie Institute of Oncology, Warsaw
- Portugal (6):
  - Centro Clinico Academico - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimaraes, Guimarães
  - Centro Hospitalar de Lisboa Central, E.P.E . - Hospital de Santo Antonio dos Capuchos, Lisbon
  - Fundacao Champalimaud, Lisbon
  - Centro Hospitalar Lisboa Norte, EPE, Lisbon
  - Unidade Local de Saude de Matosinhos EPE - Hospital Pedro Hispano, Matosinhos Municipality
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (4):
  - Wilgers Oncology Centre, Gauteng
  - Wits Clinical Research, Johannesburg
  - The Medical Oncology Centre of Rosebank, Johannesburg
  - Cape Town Oncology Trials, Kraaifontein
- South Korea (9):
  - Samsung Medical Center, Gangnam-Gu
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Gyeongsangbuk-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (19):
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario De Elche, Elche
  - Hospital Universitario de Jaen, Jaén
  - Hospital Beata María Ana, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Santiago de Compostela - CHUS, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano De Oncologia (IVO), Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (10):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (5):
  - Barts Cancer Institute, London
  - University College London Hospitals, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tarantino P, Tolaney SM, Curigliano G. Trastuzumab deruxtecan (T-DXd) in HER2-low metastatic breast cancer treatment. Ann Oncol. 2023 Oct;34(10):949-950. doi: 10.1016/j.annonc.2023.07.003. Epub 2023 Jul 26. No abstract available. PMID 37499870
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT05840211